CLINICAL TRIAL: NCT00000359
Title: Treatments for Benign Paroxysmal Positional Vertigo (BPPV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Helen Cohen, Professor, Baylor College of Medicine
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: NIDCD-1156; R01DC003602 (NIH); 1R01DC003602-01A1 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Vertigo
Keywords: Physical Therapy; Vertigo; rehabilitation; occupational therapy
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Canalith repositioning maneuver (Experimental): Repositioning treatment for posterior canal BPPV
  Interventions: Behavioral: Canalith repositioning maneuver (Epley maneuver)
- Modified Epley maneuver (Experimental)
  Interventions: Behavioral: Vestibular habituation exercises
- Sham (Sham Comparator): The subject sat in a chair; the head was passively tilted downward, turned away from the involved side, turned back to center, upward, away from the involved side, twice, slowly.
  Interventions: Behavioral: ShamManeuver
- Liberatory maneuver (Active Comparator): The standard liberatory maneuver (also known as the Semont maneuver) was used.
  Interventions: Behavioral: Semont maneuver
- Brandt Daroff exercise (Active Comparator): Modified Brandt Daroff exercise performed as a self-liberatory exercise.
  Interventions: Behavioral: Brandt-Daroff exercises

INTERVENTIONS:
Behavioral: Canalith repositioning maneuver (Epley maneuver) — Standard passive motion of the head: Dix-Hallpike maneuver, turn head to opposite side, roll over, sit up.
  Other Names: CRP; Epley maneuver
  Arms: Canalith repositioning maneuver
Behavioral: Semont maneuver — Sidelying maneuver, flip over 180 deg, sit up.
  Other Names: Liberatory maneuver
  Arms: Liberatory maneuver
Behavioral: Brandt-Daroff exercises — Active exercise. Sidelying to involved side, sidelying to uninvolved side, sit up.
  Arms: Brandt Daroff exercise
Behavioral: Vestibular habituation exercises — Head shaking exercises in pitch, roll, yaw and circumduction. Titrating from 2 repetitions per exercise to 20 repetitions per exercise, as tolerated.
  Arms: Modified Epley maneuver
Behavioral: ShamManeuver — Passive movement of the head
  Arms: Sham

SUMMARY:
The purpose of this study was to determine the relative short- and long-term efficacy of several physical treatment paradigms commonly employed for the treatment of benign paroxysmal positional vertigo (BPPV), including the canalith repositioning (Epley) maneuver, the liberatory (Semont) maneuver, the Brandt-Daroff exercises and nonspecific vestibular habituation exercises. These procedures involve exercises and head manipulations. Vertigo intensity and frequency, the presence/absence of slow-phase eye movements, the degree of dizziness handicap and acts of daily living (ADL) were assessed. The study also ascertained the effects of co-morbid conditions on the response to treatment. While BPPV is a common and significant public health problem that has been recognized for several decades, this is the first systematic study of the relative treatment efficacy of different physical treatment modalities for this disorder.

ELIGIBILITY:
Inclusion Criteria:

Patients may be eligible for this study if they:

* Are at least 21 years old.
* Have a diagnosis of unilateral posterior semicircular canal BPPV according to established clinical test criteria.
* Have functional to normal range of motion of the neck and the back.

Exclusion Criteria:

Patients will not be eligible for this study if they:

* Have a history of prior ear surgery or prior treatment for BPPV.
* Have an orthopedic or connective tissue disorder that impairs functional neck or trunk range of motion.
* Have a significant neurological disorder or spinal cord damage.
* Are on vestibular suppressant medications.
* Have Meniere's disease or acoustic neuromas.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 1998-10; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Vertigo | 6 month s

SECONDARY OUTCOMES:
Balance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Helen Cohen, EdD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Cohen HS. Side-lying as an alternative to the Dix-Hallpike test of the posterior canal. Otol Neurotol. 2004 Mar;25(2):130-4. doi: 10.1097/00129492-200403000-00008. PMID 15021771
- [Result] Cohen HS, Kimball KT, Stewart MG. Benign paroxysmal positional vertigo and comorbid conditions. ORL J Otorhinolaryngol Relat Spec. 2004;66(1):11-5. doi: 10.1159/000077227. PMID 15103195
- [Result] Cohen HS, Kimball KT. Treatment variations on the Epley maneuver for benign paroxysmal positional vertigo. Am J Otolaryngol. 2004 Jan-Feb;25(1):33-7. doi: 10.1016/j.amjoto.2003.09.010. PMID 15011204
- [Result] Cohen HS, Kimball KT. Effectiveness of treatments for benign paroxysmal positional vertigo of the posterior canal. Otol Neurotol. 2005 Sep;26(5):1034-40. doi: 10.1097/01.mao.0000185044.31276.59. PMID 16151355